CLINICAL TRIAL: NCT02782650
Title: Prenatal Counseling in Extreme Prematurity: Professionals' View
Acronym: PreCo-profs
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); UMC Utrecht (Other); Leiden University Medical Center (Other); Erasmus Medical Center (Other); Maastricht universitair medisch centrum, Maastricht (Unknown); Isala (Other); University Medical Center Groningen (Other); Maxima Medical Center (Other); Amsterdam UMC, location VUmc (Other)
Responsible Party: Sponsor
Other Study IDs: Preco-1
Record Dates: First submitted 2016-05-10; First posted 2016-05-25 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Premature Birth; Extremely Premature Infants
Keywords: Limits; Prenatal Counseling; Decision-making; Foetal Complications; Counseling; Viability
MeSH Terms: conditions — Premature Birth | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Survey and interviews: * part one * (quantitative)
  Survey on:
  A) prenatal counseling at the limits of viability, both current and preferred, within three domains of interest:
  * organization of prenatal counseling
  * content of prenatal counseling
  * decision-making in prenatal counseling
  B) treatment options at the limits of viability against the background of the Dutch guideline
  * part two * (qualitative)
  Focus groups interviews (qualitative) to in-depth explore preferences in prenatal counseling
  * insight in the specific preferred content of prenatal counseling.
  * study influencing factors on preferences in the domains of organization and decision-making.
  Interventions: Other: survey and interview

INTERVENTIONS:
Other: survey and interview — all participants: survey on prenatal counseling and treatment decisions at the limits of viability.
  a selection of participants: focus group interviews to further perform in-depth exploration of prenatal counseling preferences

SUMMARY:
This study is part of the PreCo study, evaluating Dutch care in (imminent) extreme preterm birth including current and preferred counseling, barriers and facilitators for preferred counseling from both obstetricians and neonatologists, as well as parents' views on this.

Since 2010, intensive care can be offered in the Netherlands at 24+0 weeks gestation (with parental consent) but as some international guidelines, the Dutch guideline lacks detailed recommendations on organization, content and preferred decision-making of the counseling.

DETAILED DESCRIPTION:
The anticipated delivery of an infant at the limits of viability presents parents and professionals with medical, ethical and emotional issues; especially when a decision on the initiation of care has to be made. Since the first publication in 2002 by the American Academy of Pediatrics several (albeit different) guidelines and recommendations on periviability counseling have been published. However, there is no universally accepted way of performing prenatal counseling and, consequently, studies describe heterogeneous counseling practices worldwide.

Some guidelines on resuscitation at the limits of viability include recommendations on the parental involvement in the decision-making. Nevertheless, the extent of involvement and the gestational age (GA) at which parents should be involved, varies. In 2010, the Dutch guideline on perinatal practice in extremely premature delivery lowered the limit offering intensive care from 25+0 to 24+0 weeks GA. Just as some international guidelines include a role for parents at the limits of viability, the Dutch guideline states that at 24 weeks GA informed consent of parents is required when initiating intensive care28. Although the guideline acknowledges the importance of prenatal counseling, recommendations on organization, content or decision-making of the counseling are very limited.

Although recommendations on counseling do exist, they may not be generally applicable in the Netherlands since cross-cultural differences in perinatal practices, healthcare organization, and physician and patient views are likely to exist. To compose a national framework on prenatal counseling at the limits of viability, the nationwide PreCo study (Prenatal Counseling in Prematurity) was designed, examining both professional and parental views. High quality of care originates when no differences exist between preferred and current counseling with uniformity between the involved caregivers (obstetricians and neonatologists) and specified to the needs of those receiving counseling

The PreCo study amongst professionals has three major aims

1. to find initial preferences among Dutch perinatal professionals (neonatologists and obstetricians) on prenatal counseling at the limits of viability (quantitatively)
2. to investigate Dutch physicians' preferences on decisions about treatment options for an extremely premature neonate against the background of the Dutch guideline.(quantitatively)
3. to perform in-depth exploration of counseling preferences amongst Dutch perinatal professionals (qualitatively)

ELIGIBILITY:
Inclusion Criteria:

* (fellow) neonatologist OR (fellow) obstetrician from one of the 10 specialized perinatal care centers in the Netherlands

Exclusion Criteria:

* member of the study group

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All (fellow) neonatologists OR (fellow) obstetricians from one of the 10 specialized perinatal care centers in the Netherlands
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2012-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
current and preferred prenatal counseling practices in 3 domains (organization, content, decision-making) | during the time of the survey (july 2012 - dec 2013)
preferences in treatment decisions (organization, content, decision-making) | during the time of the survey (july 2012 - dec 2013)
qualitative explored specific preferences in content, influencing factors on organization and decision-making | during focus group interviews (may - july 2015)

SECONDARY OUTCOMES:
differences between neonatologists and obstetricians | during the time of the survey (july 2012 - dec 2013)

CONTACTS AND LOCATIONS:
Overall Officials: Marije Hogeveen, MD, PhD, Principal Investigator — Radboud University Medical Center

IPD SHARING:
Plan to Share IPD: Undecided
available upon request

REFERENCES:
- [Derived] Geurtzen R, Van Heijst A, Hermens R, Scheepers H, Woiski M, Draaisma J, Hogeveen M. Preferred prenatal counselling at the limits of viability: a survey among Dutch perinatal professionals. BMC Pregnancy Childbirth. 2018 Jan 3;18(1):7. doi: 10.1186/s12884-017-1644-6. PMID 29298669